CLINICAL TRIAL: NCT06583915
Title: Comparative Study of Dry Needling Vs Transcutaneous Electrical Nerve Stimulation in Management of Patient with Myofascial Pain Dysfunction Syndrome Using Electromyography and Visual Analogue Scale: a Randomized Clinical Trial
Brief Title: Dry Needling Vs Transcutaneous Electrical Nerve Stimulation in Management of Myofascial Pain Dysfunction Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amina amr sayed mohamed salama, Master Degree Student, Department of oral and maxillofacial surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OMFS333
Record Dates: First submitted 2024-08-31; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Myofascial Pain - Dysfunction Syndrome of TMJ
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transcutaneous electrical nerve stimulation (Experimental): Low voltage electrical pulses that are applied to the central nervous system
  Interventions: Procedure: TENS
- Dry Needling (Active Comparator): insertion of a solid filiform needle into a trigger point without the administration of any substance
  Interventions: Procedure: Dry Needle

INTERVENTIONS:
Procedure: TENS — Non-pharmacological method which is widely used by medical and paramedical professionals for the management of acute and chronic pain using electric pulse generator, lead wires and electrodes.
  Arms: Transcutaneous electrical nerve stimulation
Procedure: Dry Needle — Invasive procedure where a fine needle or acupuncture needle is inserted into the skin and muscle.
  Arms: Dry Needling

SUMMARY:
Myofascial pain dysfunction syndrome (MPDS) is the most common form of temporomandibular disorders. Because of the multifactorial nature of the problem, its management is still not definite. This randomized clinical trial aimed to assess the efficacy of transcutaneous electrical nerve stimulation over dry needling for management of such condition.

DETAILED DESCRIPTION:
Myofascial pain syndrome (MPS) is a prevalent affliction among individuals experiencing musculoskeletal pain issues. This condition is characterized by pain originating from the muscle and surrounding fascia. Patients typically exhibit localized pain in a confined region or referred pain with diverse patterns.

Additionally, physical examinations may reveal trigger points on the affected muscles. MPS can be categorized into acute and chronic forms. Acute MPS often resolves spontaneously or with uncomplicated treatments. However, chronic MPS typically has a poorer prognosis, and symptoms may persist for six months or more.

Dry needling involves the insertion of a solid filiform needle into a trigger point without the administration of any substance. Various theories have been put forth to explain the mechanisms by which dry needling alleviates pain . These include the "gate control" theory, modulation of endogenous opioids such as B-endorphin, encephalins, and dynorphins, disruption of central sensitization through activation of Aβ fibers resulting in inhibition of synaptic transmission between Aβ and C fibers and cells of the spinal cord dorsal horn due to their slower impulse conduction, and even placebo effects have been suggested . When a needle is inserted into a trigger point, it may elicit a local twitch response. This reflexive contraction of the trigger point can also facilitate physiological changes, including the reduction of spontaneous electrical activity and the concentration of inflammatory and nociceptive chemicals, ultimately resulting in the relaxation of the trigger point.

Transcutaneous electrical nerve stimulation (TENS) is considered to be a highly secure and cost-effective modality for managing both chronic and acute pain. As per the gate control theory, TENS employs low voltage electrical pulses that are applied to the central nervous system. The modulation of pain perception induced by TENS is attributed to the recruitment of Aβ afferent fibers in the posterior horn of the spinal cord, which prevents the activation of pain conducted in thin fiber. Electrical stimulation effectively inhibits the transmission of painful impulses through the spinal cord and stimulates the release of endogenous opioids by the brain. Its safe, noninvasive, inexpensive and effective method of providing analgesia with reduced potential adverse effects compared to other treatment modalities.

In this research, we aim to evaluate TENS is a suitable treatment for MPDS patients, which would eliminate the need for another treatment modality. The expected benefit in this study is to find the best treatment for MPDS reducing pain, muscle stiffness and limited mouth opening.

ELIGIBILITY:
Inclusion Criteria:

1. Patients complaining of pain in muscles of mastication lasting for three months or more.
2. Presence of trigger points in the temporalis, masseter or lateral pterygoid muscle identified by clinical examination and palpation.
3. Average pain severity of at least 4 on a 10-point scale
4. Pain in pre-auricular area, or in the ear during rest or function

Exclusion Criteria:

1. No previous tempro-mandibular joint (TMJ) surgical intervention
2. Patients with neurological disorders, coagulopathy, vascular disease autoimmune disease (systemic lupus, rheumatoid arthritis), fibromyalgia
3. Pregnancy
4. Current opioid use
5. Intake of analgesics, muscle relaxant, anti-inflammatory medications such as NSAID's and benzodiazepines,
6. Patients with severe trauma or infections in TMJ
7. Tempro-mandibular dysfunction (TMD) with joint origin (any type of internal derangement)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Pain | From enrollment to the end of treatment at 6 months
  Using visual analogue scale (VAS) from (1-10) where 1 is the least pain and 10 is the maximum pain

SECONDARY OUTCOMES:
Muscle stiffness | From enrollment to the end of treatment at 6 months
  using Electromyography to measure muscle response or electrical activity in response to a nerve stimulation of the muscle (volt)
Limitation in mouth openinig | From enrollment to the end of treatment at 6 months
  Measuring muscle opening using digital caliber (Micrometer)
Sleeping disorder | From enrollment to the end of treatment at 6 months
  Assessing sleeping disorder through Yes or No questionnaire
Anxiety | From enrollment to the end of treatment at 6 months
  Assessing anxiety through Yes or No questionnaire
Patient satisfaction | From enrollment to the end of treatment at 6 months
  Assessing patient satisfaction through Yes or No questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa ElGengehy, PhD, Study Chair — Professor, Department of oral and maxillofacial surgery

IPD SHARING:
Plan to Share IPD: No
lack of research ethics committee approval of secondary use of IPD